CLINICAL TRIAL: NCT07155759
Title: Long-term Outcomes of Prostate Cancer Screening Using PSA, Biomarkers and MRI: The STHLM3MRI Trial
Brief Title: Long-term Outcomes of Prostate Cancer Screening
Acronym: STHLM3MRI_3
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Swedish Cancer Foundation (Other); The Swedish Research Council (Other Government)
Responsible Party: Principal Investigator, Tobias Nordström, Associate Professor, Consultant Urologist, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: STHLM3MRI_3
Record Dates: First submitted 2025-08-20; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer
Keywords: screening; magnetic resonance imaging; biomarker; mortality; stockholm3
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes are verified through national registers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Organized screening including repeat testing (MRI+biomarkers) (Experimental): participants are offered prostate cancer screening. Interventions are (i) a paired PSA and Stockholm3 bloodtest; (ii) if elevated (PSA>=3 | Stockholm3>=0.11), an MRI is offered. If MRI shows PI-RADS≥3, prostate biopsies are offered. Screenings are offered at year 0, year 2-3 (if original PSA≥1.5) and year 6
  Interventions: Diagnostic Test: PSA/Stockholm3/MRI
- One-time invitation to testing arm (traditional biopsies) (Active Comparator): participants are offered prostate cancer screening. interventions are a PSA bloodtest. If PSA≥3 ng/ml, a standard prostate biopsy is offered. No repeat screenings are offered.
  Interventions: Diagnostic Test: PSA
- Population controls (No Intervention): Population controls are identified through registers and followed in national outcome registers (Swedish Board of Health and Welfare)

INTERVENTIONS:
Diagnostic Test: PSA/Stockholm3/MRI — Stockholm3+PSA followed by MRI of the prostate
  Arms: Organized screening including repeat testing (MRI+biomarkers)
Diagnostic Test: PSA — PSA followed by standard biopsies
  Arms: One-time invitation to testing arm (traditional biopsies)

SUMMARY:
This study is an expansion of the screening-by-invitation STHLM3MRI trial for detection of prostate cancer. In summary, we assess longterm outcomes (prostate cancer mortality, incidence and resource use) in men (i) invited and randomized to a screening program using PSA, a biomarker test and MRI; (ii) invited and randomized to a single PSA test with prostate biopsies followed by opportunistic testing and (iii) population controls. Mortality is verified through register data, disease verification is made through in-study biopsy results and registry data.

ELIGIBILITY:
Eligible participants:

-Men eligible for the longterm f/u-study arms (experimental and control) are participants in the STHLM3MRI trial.

Inclusion Criteria:

* Men age 50-74 years without prior diagnosis of prostate cancer (ICD-9 C61).
* Permanent postal address in Stockholm
* Not a previous participant in the Stockholm3 study (2012-2014)

Exclusion Criteria:

* Severe illnesses such as metastatic cancers, severe cardio-vascular disease or dementia
* Contraindications for magnetic resonance imaging (MRI) eg pacemaker, magnetic cerebral clips, cochlear implants or severe claustrophobia.
* Men with a previous prostate biopsy the preceding 60 days before invitation.

Ages: 50 Years to 74 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7500 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2035-11 (Estimated)

PRIMARY OUTCOMES:
Prostate cancer mortality | 5-10 years
  Mortality from prostate cancer (yes/no)
Detection of clinically significant prostate cancer | 1-3 years
  Gleason Score ≥7 disease detected (Yes/No)

SECONDARY OUTCOMES:
Prostate cancer metastasis-free survival | 5-10 years
Detection of prostate cancer by grade | 1-3 years
  ISUP (International Society of UroPathology) grade group 1-5
Performed prostate biopsy | 1-3 years
  Participant undergone a biopsy procedure of the prostate (Yes/No)
Performed MRI of prostate | 1-3 years
Grading of MRI prostate | 1-3 years
  PI-RADS (Prostate Imaging Reporting and Data System (PI-RADS)
  ) score (1-5)

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Nordström, Ass Prof, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data underlying the results reported in this project will be available after deidentification, together with the study protocol, statistical analysis plan, and analytic code. Data will be made available to researchers who provide a methodologically robust proposal, in which the aims are relevant and clear. Proposals can be submitted up to 24 months after publication of the first main article of the project and should be directed to tobias.nordstrom@ki.se. Only proposals with ethical approval will be granted access to the data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 24 months from publication of first main manuscript of the project